CLINICAL TRIAL: NCT07298538
Title: Long-term Survival of Unresectable Hepatocellular Carcinoma Patients Receiving Lenvatinib-based Therapy: A Retrospective, Multicenter Propensity Score Matching Study
Brief Title: Long-Term Survival With Lenvatinib-Based Therapy in Unresectable Liver Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: bc20254383
Record Dates: First submitted 2025-11-25; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Unresectable Hepatocellular Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lenvatinib-based therapy
- Non-lenvatinib therapy

SUMMARY:
This study reviewed real-world outcomes of patients with unresectable hepatocellular carcinoma who received lenvatinib-based treatment. The study evaluated long-term survival, treatment response, and safety using data collected from six hospitals.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Patients with histologically or radiologically confirmed HCC who were newly diagnosed between January 2019 and December 2022 (meeting the diagnostic criteria of the American Association for the Study of Liver Diseases or the Chinese Guidelines for the Diagnosis and Treatment of Primary Liver Cancer).
* Patients with at least 1 measurable lesion in the liver per RECIST v.1.1.
* Initially unresectable HCC as determined by the investigator (including oncologically unresectable, surgically unresectable, or both).
* Child Pugh score ≤ 7
* ECOG-PS 0-1
* Patients who had not received any previous systemic therapy before receiving dual therapy (lenvatinib + immunotherapy/local therapy) or triple therapy (lenvatinib + immunotherapy + local therapy) as the first-line therapy. Combination therapy is defined as the initiation of immunotherapy or local therapy within 30 days (before or after) of the first dose of lenvatinib.
* Patients who had basic image data (CT/MRI/PET) and underwent at least one imaging evaluation during the systemic therapy (if the image data was obtained from other hospitals, the original data shall be provided for re-evaluation).

Exclusion Criteria:

* Patients with no overall survival (OS) endpoint observed, and a follow-up period after treatment initiation of less than 6 months.
* Patients with a pathological diagnosis of combined hepatocellular and intrahepatic cholangiocarcinoma (cHCC-ICC), cholangiocarcinoma, or other non-HCC malignant tumors.
* Patients with other inadequately treated malignant tumors previously or currently.
* Prior liver transplantation/hepatectomy/ablation for liver cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unresectable Hepatocellular Carcinoma Patients Receiving Lenvatinib-based Therapy
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
3-year Overall Survival Rate Estimated by Kaplan-Meier Method | 3 years after treatment initiation
  3-year cumulative survival rate estimated based on the Kaplan-Meier method

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 5 years after treatment initiation
  The time interval from treatment initiation to the date of death due to any cause
Event-free survival (EFS) | Up to 5 years after treatment initiation
  The time interval from treatment initiation to the occurrence of any event, including disease progression, recurrence (surgical patients), discontinuation of treatment for any reason, or death. EFS is assessed by RECIST v1.1.
4-year and 5-year OS rates | 4 years and 5 years after treatment initiation
  4-year and 5-year cumulative survival rates estimated based on the Kaplan-Meier method
Objective response rate (ORR) | Up to 12 months after treatment initiation
  The proportion of patients who achieved the best overall response (BOR) of complete response (CR) or partial response (PR) as assessed by the investigator per RECIST v1.1
Incidence of Adverse Events (AEs) and Surgical Complications | AEs: from treatment initiation through 30 days after last dose of lenvatinib-based therapy; Surgical complications: perioperative period (day of surgery through 30 days post-surgery)
  Adverse Events and surgical complications

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China